CLINICAL TRIAL: NCT06911918
Title: The Effect of Time Restricted Eating on Glycemic and Proinflammatory Biomarkers Among Prediabetic Obese Jordanian Adults Aged 18-40 Years Old: A Randomized Control Study
Brief Title: The Effect of Time Restricted Eating on Glycemic and Proinflammatory Biomarkers Among Prediabetic Obese Jordanian Adults Aged 18-40 Years Old
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Najd AlSarayreh, Principal investigator, PhD Candidate in Human Nutrition and Dietetics, University of Jordan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 382/2025
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Insulin Resistance; Inflammation Biomarkers; Time Restricted Eating; Caloric Restriction; Obesity (Disorder)
Keywords: Time restricted eating; Insulin Resistance; Obesity; Caloric Restriction; Inflammation cytokines
MeSH Terms: conditions — Insulin Resistance; Intermittent Fasting; Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: This open-label, 12-week randomized controlled experimental trial factorial 2X2 with a 1:1 allocation ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 10-h Time restricted eating with caloric restriction (Experimental)
  Interventions: Other: time restricted eating with caloric restriction
- 10-h time restricted eating without caloric restriction (Active Comparator)
  Interventions: Other: time restricted eating without caloric restriction
- caloric restriction without time restricted eating (Active Comparator)
  Interventions: Other: Caloric restriction without Time restricted eating
- No time restricted eating - normal diet (Active Comparator)
  Interventions: Other: No time restricted eating - Normal diet

INTERVENTIONS:
Other: time restricted eating with caloric restriction — will be asked to reduce their energy intake by 550 each day. Total energy expenditure will be calculated using the Bioelectrical impedance (BIA); Inbody 120 and multiplied by the physical activity factor and reduced by 550 kilo calories for each participant. The acceptable macronutrient distribution range (AMDR) will be 45-60% carbohydrates, 15-25% protein, and 20-30% fat of the total caloric value and fasted from 18:00 to 8:00 daily (a 14-h fast) in the 12-weeks intervention
  Arms: 10-h Time restricted eating with caloric restriction
Other: time restricted eating without caloric restriction — will be asked to maintain their normal diet to the acceptable normal distribution ranges and fast from 8:00 to 18:00. They do not need to restrict caloric intake during the feeding window
  Arms: 10-h time restricted eating without caloric restriction
Other: Caloric restriction without Time restricted eating — will be asked to reduce their energy intake by 550 each day. Total energy expenditure will be calculated using the Bioelectrical impedance (BIA); Inbody 120 and multiplied by the physical activity factor and reduced by 550 kilo calories for each participant. The acceptable macronutrient distribution range (AMDR) will be 45-60% carbohydrates, 15-25% protein, and 20-30% fat of the total caloric value
  Arms: caloric restriction without time restricted eating
Other: No time restricted eating - Normal diet — will be asked to maintain their normal diet as the second intervention arm without time restricted eating throughout the trial
  Arms: No time restricted eating - normal diet

SUMMARY:
Obesity, a global epidemic, significantly contributes to prediabetes, cardiovascular diseases, and other chronic diseases due to its pro-inflammatory nature. This studyl investigates the effects of time-restricted eating (TRE) with calorie restriction (CR), TRE without CR, and CR without TRE on glycemic control and pro-inflammatory biomarkers among prediabetic obese Jordanian adults aged 18-40 years. The study assesses changes in pro-inflammatory biomarkers (IL-1β, TNF-α, IL-6), insulin resistance (HOMA-IR), and body composition over 12 weeks.

Participants (n=120) will be randomized into four intervention arms: (1) TRE with CR, (2) TRE without CR, (3) CR without TRE, and (4) a control group with no dietary restrictions and no TRE. Biweekly anthropometric assessments will evaluate pro-inflammatory biomarkers and biochemical measures at baseline and the end of the study. The findings will provide insights into the comparative effectiveness of TRE and CR, potentially offering a safe, cost-effective intervention to prevent obesity-induced inflammation, prediabetes, and progression to type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* IR individuals diagnosed with IR by the physicians as indicated by HOMA-IR score
* female and male, BMI ≥ 30 to 39.9 kg/m2
* age between 18 and 40 years
* stable weight for 3 months before the beginning of the study
* sedentary lifestyle

Exclusion Criteria:

* previous weight loss surgery
* pregnancy or intent to become pregnant
* breastfeeding
* chronic diseases
* drug therapies that could interfere with the effectiveness of the dietary intervention (e.g., use of corticosteroids, and anti-diabetic drugs)
* diabetic type 1 and 2 individuals
* anyone physically active to reduce the influence of confounding covariates

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Serum of TNF-α, IL-1β and IL-6 | baseline and after 12 weeks of intervention
  Will be measured using ELISA before and after dietary intervention to assess the impact of time restricted eating on these proinflammatory biomarkers in participants diagnosed with Insulin resistance

SECONDARY OUTCOMES:
Homa-IR | baseline and after 12 weeks of intervention
  Homa-IR will be assessed using the homeostasis model assessment (HOMA) method, which involves applying the formula [fasting glucose (mg/dL) * fasting insulin (mU/mL)/ 405] to evaluate the changes in insulin resistance over 12 weeks of intervention
Lipid profile (LDL, HDL, TG, and cholesterol) | baseline and after 12 weeks of intervention
  will be analyzed at based line and post intervention to determine the impact of dietary modification on lipid profile
body weight | baseline and every 2 weeks until 12 weeks of intervention
  in kilograms (Using inbody 120 )
Dietary intake using food records | week4, week 8, and week 12 week
Fasting blood glucose | baseline and after 12 weeks of intervention
fasting insulin level | baseline and after 12 weeks of intervention
height | baseline
  in centimeters, Height measuring scale - Stadiometer without shoes
Body composition | baseline and every 2 weeks until 12 weeks of intervention
  %fat, fat in kilo grams, muscle mass in kilograms, using inbody 120

CONTACTS AND LOCATIONS:
Locations (1):
- Najd Nutri Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The individual participant data IPD will not be shared due to privacy concerns and institutional polices. Data access is restricted to the research team to ensure confidentially and compliance with ethical guidelines